CLINICAL TRIAL: NCT00365833
Title: Circulating Endothelial Cell and Endothelial Progenitor Cell Evaluation of Kidney Transplant Patients
Brief Title: CEC/EPC and Cardiovascular Risk in Renal Transplant Recipients
Acronym: CEC
Status: Terminated | Type: Observational
Why Stopped: difficulty obtaining required data
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: 217-2006
Record Dates: First submitted 2006-08-17; First posted 2006-08-18 (Estimated); Last update posted 2011-09-30 (Estimated); Status verified 2011-09

CONDITIONS: Transplantation, Kidney; Cardiovascular Abnormalities; Cardiovascular Diseases
Keywords: Transplantation; Cardiovascular; Renal
MeSH Terms: conditions — Cardiovascular Abnormalities; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Recipients of Kidney Transplant: Patients Transplanted with Live or Deceased Donor's Kidney. Standard of Care treatment pre- and post-transplant.

SUMMARY:
We believe that certain cells in the human body (Circulating Endothelial Cells and Endothelial Progenitor Cells) are related to risk of cardiovascular disease. It may be possible to measure levels of these cells in patients who have had a kidney transplant and predict their risk of developing cardiovascular disease.

DETAILED DESCRIPTION:
Coronary disease is one of the most common causes of morbidity and mortality in patients with known chronic renal insufficiency and those with end stage renal disease. Consequently, early detection with markers such as circulating endothelial cells and endothelial progenitor cells has been studied in order to identify vascular function and assess overall cardiovascular risk. Based on current research, there exists a notable increase in Circulating Endothelial Cells (CEC) and a reduction of Endothelial Progenitor Cells (EPC) with renal dysfunction due to endothelial damage. Therefore circulating endothelial cells are a marker for cardiovascular health.

Renal transplant patients also possess a higher cardiovascular risk than the general population, but have known improvement in survival as compared to patients with ESRD (End Stage Renal Disease). In addition, because of the excellent outcomes, graft and patient survival and even acute rejection are no longer very useful endpoints for clinical studies. The tolerability of transplant drug regimens and the impact of these regimes on cardiovascular health in kidney transplantation has become, consequently, a new focus of research. Currently, no clear long-term analysis has been fulfilled analyzing CEC or EPC in this group of patients. We hypothesize that CEC can serve as biological markers for cardiovascular risk assessment in cadaveric and living renal transplant patients. We eventually hope measurement of these cells can serve as an endpoint in determining cardiovascular outcome in renal transplant patients. Our present study is aimed to get an initial assessment of the kinetics of CEC and EPC in renal transplant recipients just prior to transplant and for the first two years post transplant.

ELIGIBILITY:
Inclusion Criteria:

* kidney transplant recipients
* kidney/pancreas transplant recipients
* age 18-80

Exclusion Criteria:

* inability to return for follow-up visits
* multiple organ transplant other than listed above

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: de novo renal transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2006-07; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Cardiovascular Risk Profile | 24 months
  Cardiovascular Risk Profile is defined by calculated Framingham Model

SECONDARY OUTCOMES:
Rate of Cardiovascular Events Post-Transplant | 24 months
  Measured by Kaplan-Meier analysis and Cox Proportional Hazard Models to correlate CEC and EPC to this outcome.
Rate of Patient Survival Post-Transplant | 24 months
  Measured by Kaplan-Meier analysis and Cox Proportional Hazard Models to correlate CEC and EPC to this outcome.
Rate of Graft Survival Post-Transplant | 24 months
  Measured by Kaplan-Meier analysis and Cox Proportional Hazard Models to correlate CEC and EPC to this outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Herwig-Ulf Meier-Kriesche, md, Principal Investigator — University of Florida; Giselle Guerra, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States